CLINICAL TRIAL: NCT06738875
Title: Monitoring Changes in Endotracheal Tube Cuff Pressure During Laparoscopic Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hülya Tosun Söner, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: HTONER
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Prospective Observational Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: manometre — Increases in peak and mean airway pressures of ETT cuff pressures will be monitored in patients undergoing laparoscopic bariatric surgery

SUMMARY:
This prospective observational cohort study was designed to assess the relationship between ETT cuff pressures and airway pressures in obese patients undergoing laparoscopic bariatric surgery. We hypothesized that the ETT cuff pressures will rise in direct relationship to increases in the peak and mean airway pressures.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) risk indicators I-III manage to undergo Laparoscopic bariatric surgery between the ages of 18-70

Exclusion Criteria:

* Patients with drug allergies, chronic pain, long-term opioid use, history of psychiatric illness, and need for emergency surgery were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 28
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
ETT cuff pressure | 1-immediately after intubation; 2-after intraperitoneal insufflation; 3-after the position is given 4-after peritoneal exsufflation
  ETT cuff pressure

SECONDARY OUTCOMES:
Peak airway pressures | 1-immediately after intubation; 2-after intraperitoneal insufflation; 3-after the position is given 4-after peritoneal exsufflation
  Peak airway pressures

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital, Kayapınar, Di̇yarbakir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No